CLINICAL TRIAL: NCT06642480
Title: Determination of Patients' Visual Analogue Scale (VAS) in Postoperative Patients Receiving Tramadol Analgesia in the Minangkabau Ethnic Group, Indonesia
Brief Title: Distribution of CYP2D6 Multiplication, CYP2D6*5, and Clinical Implications in Postoperative Patients Receiving Tramadol Analgesia in the Minangkabau Ethnic Group, Indonesia
Acronym: Tramadol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia (Other Government)
Collaborators: Andalas University (Other)
Responsible Party: Principal Investigator, Desriani Desriani, DR, Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BRIN; 2/III/HK/2022 (Other Grant/Funding Number: BRIN)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Post Operative Analgesia; Tramadol
Keywords: Tramadol; Post Operative; Minangkabau

STUDY DESIGN:
Intervention Model Description: VAS of 63 patients was determined by injecting tramadol at a dose of 100 mg 30 minutes before the operation was completed. It was observed in the recovery room at 30, 60, and 120 minutes. Tramadol had an onset time of 15-60 minutes, with peak effectiveness at 2-6 hours postoperatively. Pain level was categorized into 0 (no pain), 1-3 (signifying mild), 4-6 (middle), and 7-10 ( heavy pain).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Determination of Patients' Visual Analogue Scale (VAS) (Other): Pain level was categorized into 0 (no pain), 1-3 (signifying mild), 4-6 (middle), and 7-10 ( heavy pain).
  Interventions: Drug: Post Operative Analgesia

INTERVENTIONS:
Drug: Post Operative Analgesia — administering 100 mg of intravenous tramadol 30 minutes before the operation is completed
Drug: Post Operative Analgesia — VAS of 63 patients was determined by injecting tramadol at a dose of 100 mg 30 minutes before the operation was completed. It was observed in the recovery room at 30, 60, and 120 minutes.

SUMMARY:
Cytochrome P450 2D6 (CYP2D6) is an important enzyme in metabolizing commonly used drugs such as Tramadol hydrochloride (widely used opioid analgesic). Genetic polymorphisms of the CYP2D6 gene have been shown to influence the pharmacodynamic properties of the administered drug. This study aimed to screen 63 postoperative patients (wild-type, CYP2D6*5, and CYP2D6 multiplication) of Minangkabau ethnicity in West Sumatera, Indonesia, who received tramadol using a modified long PCR method and to investigate the clinical impact of tramadol on the patients.

DETAILED DESCRIPTION:
VAS of 63 patients was determined by injecting tramadol at a dose of 100 mg 30 minutes before the operation was completed. It was observed in the recovery room at 30, 60, and 120 minutes. Tramadol had an onset time of 15-60 minutes, with peak effectiveness at 2-6 hours postoperatively. Pain level was categorized into 0 (no pain), 1-3 (signifying mild), 4-6 (middle), and 7-10 ( heavy pain).

ELIGIBILITY:
Inclusion Criteria:

* Post operative patients who get analgesic tramadol

Exclusion Criteria:

* No exclusion criteria

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Determination of Patients' Visual Analogue Scale (VAS) | . It was observed in the recovery room at 30, 60, and 120 minutes
  Pain level was categorized into 0 (no pain), 1-3 (signifying mild), 4-6 (middle), and 7-10 ( heavy pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Rsup Dr M Djamil Padang, Padang, West Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Effendi R, Rizqia Haz A, Muhammad Fuad A, Dermawan B, Utami N, Desriani. Distribution of CYP2D6 multiplication, CYP2D6*5, and clinical implications in postoperative patients receiving tramadol analgesia in the Minangkabau ethnic group, Indonesia. F1000Res. 2025 Sep 23;13:1526. doi: 10.12688/f1000research.155988.3. eCollection 2024. PMID 41078883